CLINICAL TRIAL: NCT03146312
Title: Effect of a Multivitamin/Multimineral/Phytochemical Dietary Supplement on Gene Expression, Epigenetics and Nutritional Status in Healthy Adults
Brief Title: Effect of a Multivitamin/Multimineral/Phytochemical Dietary Supplement on Indices of Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USANA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 201773
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: gene expression; gene array; epigenetics; DNA methylation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVM/phytochemical supplement (Experimental): a multi-vitamin, multi-mineral, phytochemical supplement
  Interventions: Dietary Supplement: MVM/phytochemical supplement
- Placebo (Placebo Comparator): a placebo tablet (microcrystalline cellulose) identical in size, shape and color to the treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MVM/phytochemical supplement — Consumption of an MVM/phytochemical supplement for 4 weeks
  Arms: MVM/phytochemical supplement
Dietary Supplement: Placebo — Consumption of a placebo tablet identical in size, shape and color to the treatment tablet
  Arms: Placebo

SUMMARY:
This is a global transcriptomics and epigenetic pilot study designed to identify changes in gene expression and DNA methylation patterns following the consumption of an MVM/phytochemical supplement in a small group of healthy subjects. We hypothesize that genome-wide transcriptional and epigenetic studies will elucidate the molecular mechanisms underlying the health benefits associated with MVM/phytochemical supplementation.

DETAILED DESCRIPTION:
There is considerable controversy regarding the benefit of widespread dietary supplement use, in particular widespread MVM use. The controversy persists because of a marked incongruity in nutrition research: on one hand, many studies indicate that MVM supplement consumption yields few - if any - demonstrable health benefits, yet on the other hand, numerous findings indicate most Americans do not consume the RDA of a variety of nutrients, particularly vitamins and minerals, and are becoming increasingly under-nourished. Nutrigenomics offers a unique opportunity to address this controversy, as it can identify subtle changes in gene expression and epigenetic signatures immediately following a nutritional intervention - changes which may be indicative of improved health status and which may otherwise remain undetectable through other clinical endpoints for a considerable period of time, even into future generations.

Hypothesis: The investigators hypothesize that MVM/phytochemical supplementation will result in transcriptional and epigenetic changes consistent with an enhancement in human health status. Moreover, the investigators hypothesize that MVM/phytochemical supplementation will alter markers of cardiovascular, antioxidant, nutritional as well as inflammatory status in a manner indicative of improved health.

Study Design:

This will be a randomized, double blind, placebo controlled, parallel arm design conducted over a 4-week period. 50-60 healthy subjects will be recruited and, if eligible for the study, matched by age, sex and ethnicity and randomized in a 1:1 ratio to either of two interventions:

1. Daily consumption of the control supplement (placebo)
2. Daily consumption of the MVM/phytochemical supplement (treatment)

Methods:

Blood will be collected at baseline and after the 4-week intervention. At each time point, PBMCs will be collected, and DNA and RNA extracted for genome-wide gene expression and DNA methylation analyses. Serum and plasma will also be collected in order to assess clinical markers related to cardiovascular, nutritional, antioxidant and inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed Informed Consent prior to entry in the study.
* Are in generally good health.
* Comprehensive Metabolic Panel results reported within normal reference ranges
* Body Mass Index of 18.5 - 30.
* Systolic blood pressure of 90-130 mm Hg; diastolic blood pressure of 60-90 mm Hg.
* Fasting blood glucose from 65-110 mg/dl.
* Total cholesterol level of <240 mg/dl
* LDL cholesterol of <130 mg/dl
* Triglyceride level of <150 mg/dl.
* Have good venous access.
* Must be able to swallow tablets and pills

Exclusion Criteria:

* Pregnant, trying to become pregnant, or breast feeding.
* Chronic or acute use of prescription or OTC medications that may interfere with absorption of the test supplement.
* Consumption of a multivitamin/mineral or other dietary supplement for more than 5 days within 30 days of the screening visit.
* Gastrointestinal conditions that may affect consumption of the treatment or placebo tablets.
* insulin-dependent and orally controlled diabetics
* Scheduling difficulties or lack of transportation
* Have participated as a subject in any other clinical study within 30 days of the screening visit
* A history of alcohol or substance abuse within 2 years
* Significant constipation or diarrhea
* Allergies or intolerance to turmeric, curcumin or related products
* Inability or difficulty swallowing tablets and pills

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Gene expression | 4 weeks
  Gene expression measured by microarray

SECONDARY OUTCOMES:
Inflammation | 4 weeks
  change in inflammatory markers between MVM/Phytochemical Supplement and placebo
Cardiovascular Health | 4 weeks
  change in markers of cardiovascular health between MVM/Phytochemical Supplement and placebo
Nutritional status | 4 weeks
  change in markers of nutritional status between MVM/Phytochemical Supplement and placebo
Oxidative stress/Antioxidant Status | 4 weeks
  change in oxidative stress markers between MVM/Phytochemical Supplement and placebo
Epigenetics | 4 weeks
  Changes in DNA methylation patterns

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levy, PhD, Principal Investigator — USANA Health Sciences
Locations (1):
- USANA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided